CLINICAL TRIAL: NCT00693823
Title: A Prospective Randomized Comparison of Prosthetic Femoropopliteal Bypass Versus Viabahn Endoprosthesis for Treatment of Symptomatic Superficial Femoral Artery Occlusion
Brief Title: Comparison of Prosthetic Femoropopliteal Bypass Versus Viabahn Endoprosthesis for Treatment of Symptomatic Femoral Artery Occlusive Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Vascular Associates (Other)
Collaborators: W.L.Gore & Associates (Industry)
Responsible Party: Dennis R. Gable, M.D., Texas Vascular Associates/Baylor University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 003-179, Viabahn #1
Record Dates: First submitted 2008-06-03; First posted 2008-06-09 (Estimated); Last update posted 2008-06-09 (Estimated); Status verified 2008-06

CONDITIONS: Atherosclerosis; Lower Extremity Ischemia; Claudication; Rest Pain
Keywords: atherosclerosis; stent; angioplasty; covered stent
MeSH Terms: conditions — Atherosclerosis; Intermittent Claudication | interventions — Angioplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Femoral-popliteal surgical bypass with prosthetic graft
  Interventions: Procedure: Femoral-popliteal Bypass
- 2 (Active Comparator): Interventional angioplasty and placement of an ePTFE covered stent graft within the femoral-popliteal artery as an endoluminal bypass percutaneously
  Interventions: Device: Angioplasty and stent placement with Viabahn covered stent-graft(W.L. Gore & Associates, Flagstff, Arizona) of superficial femoral artery

INTERVENTIONS:
Procedure: Femoral-popliteal Bypass — Surgical placement of a prosthetic graft in the thigh from the groin to the knee
  Arms: 1
Device: Angioplasty and stent placement with Viabahn covered stent-graft(W.L. Gore & Associates, Flagstff, Arizona) of superficial femoral artery — Placement of an ePTFE covered stent graft within the superficial femoral artery in the thigh through a needle hole percutaneously
  Other Names: Viabahn endoprosthesis
  Arms: 2

SUMMARY:
This study is a comparison of two different ways to treat blockage in the artery of the thigh. The first is an older way with incisions in the groin and just above the knee. A plastic tube is then inserted to make a bypass from the groin to the knee. The second treatment offered is through a needle hole in the groin. A thin plastic tube covering a metal stent is inserted into the artery and released to bypass the blockage from inside the artery. No incisions are needed. Patients are enrolled and then selected for one treatment method or another by chance. The patients will be followed for two years to see how the two different treatment methods work compared to each other.

ELIGIBILITY:
Inclusion Criteria:Patients that had atherosclerotic stenotic or occlusive lesions of the superficial femoral artery with no significant aorto-iliac disease. The infra-popliteal segment had to be patent with at least single vessel run-off to the ankle. Patients had to be acceptable surgical candidates in the event they were randomized to the surgical arm.

-

Exclusion Criteria:Non-operative candidate,Contraindication to IV contrast use, Planned surgery with venous conduit, previously stented segment of the superficial femoral artery, poorly compliant patient.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2003-09; Primary Completion 2007-05 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Primary artery/graft patency | 24 months
Limb Salvage | 24 months
Improvement in symptoms of lower extremity Ischemia | 24 Months

SECONDARY OUTCOMES:
Secondary artery/graft patency | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States

REFERENCES:
- [Background] Lammer J, Dake MD, Bleyn J, Katzen BT, Cejna M, Piquet P, Becker GJ, Settlage RA. Peripheral arterial obstruction: prospective study of treatment with a transluminally placed self-expanding stent-graft. International Trial Study Group. Radiology. 2000 Oct;217(1):95-104. doi: 10.1148/radiology.217.1.r00se0595. PMID 11012429
- [Background] Hartung O, Otero A, Dubuc M, Boufi M, Barthelemy P, Aissi K, Alimi YS. Efficacy of Hemobahn in the treatment of superficial femoral artery lesions in patients with acute or critical ischemia: a comparative study with claudicants. Eur J Vasc Endovasc Surg. 2005 Sep;30(3):300-6. doi: 10.1016/j.ejvs.2005.04.027. PMID 15936230
- [Background] Fischer M, Schwabe C, Schulte KL. Value of the hemobahn/viabahn endoprosthesis in the treatment of long chronic lesions of the superficial femoral artery: 6 years of experience. J Endovasc Ther. 2006 Jun;13(3):281-90. doi: 10.1583/05-1799.1. PMID 16784314